CLINICAL TRIAL: NCT05482516
Title: Evaluating Novel Therapies and ctDNA as a Marker in Curatively-Treated Gastrointestinal Cancers With Microscopic Residual Disease
Brief Title: Evaluating Novel Therapies in ctDNA Positive GI Cancers
Acronym: MRD-GI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Genentech, Inc. (Industry); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005282; ML43975 (Other: Funding source)
Record Dates: First submitted 2022-07-26; First posted 2022-08-01 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Colon Adenocarcinoma; Rectal Adenocarcinoma; Gastric Adenocarcinoma; Pancreatic Adenocarcinoma; Hepatocellular Carcinoma; Adenocarcinoma of Biliary Tract; Gallbladder Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab plus Bevacizumab (Experimental): atezolizumab 1200 mg and bevacizumab 15 mg/kg given intravenously on Day 1 of each 21-day cycle (every 3 weeks [Q3W]) for a maximum of 12 months.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a monoclonal antibody that belongs to a class of drugs that bind to either the programmed death-receptor 1 (PD-1) or the PD-ligand 1 (PD-L1), blocking the PD-1/PD-L1 pathway,
  Other Names: TECENTRIQ
Drug: Bevacizumab — Bevacizumab is a tumor-starving (anti-angiogenic) therapy. Avastin is designed to block a protein called vascular endothelial growth factor, or VEGF.
  Other Names: Avastin

SUMMARY:
This study is a non-randomized, open-label, multi-cohort, multi-site, pilot feasibility therapeutic trial. The study will enroll 20 patients across 4 cohorts (CRC, gastric, PDAC, and HCC/intra-hepatic-/extra-hepatic-, gall bladder adenocarcinomas) diagnosed with histologically confirmed GI cancers. These patients will have already completed all Standard of Care (SOC) treatments (including neoadjuvant, surgery, local therapies, and/or adjuvant therapy as applicable), as defined by the treating primary physician or research team, with curative intent but have a positive SignateraTM tumor-informed ctDNA test and NED radiographically by standard imaging within 28 days prior to enrollment and within 1 year of completing all curative-intent therapy. All patients will be treated with intravenous (IV) atezolizumab 1200 mg IV and bevacizumab 15 mg/kg on Day 1 of 21-day cycles until disease recurrence, ctDNA POD, unacceptable toxicity, or subject withdrawal of consent with a maximum 12 month total duration of study therapy. Atezolizumab and bevacizumab drug will be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Age >= 18 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol, in the investigator's judgment
4. Histologically or cytologically confirmed colorectal adenocarcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, hepatocellular carcinoma, or extra-hepatic/intra-hepatic/gallbladder adenocarcinoma. Patients may be enrolled irrespective of any mutational analyses.
5. Must have been diagnosed with any stage disease (including localized and metastatic disease) that was felt to have already been treated completely with curative-intent per investigator's, primary physician's, or research team's judgement. Curative-intent treatment strategies are unique to each tumor type and stage but includes all surgeries and perioperative therapies recommended. If patients were appropriately treated with curative intent but felt to be high-risk for relapse, they may be still be included.

   o Patients diagnosed with hepatocellular carcinoma specifically must have Child Pugh A score at the time of screening; o Patients must have completed all definitive SOC treatment with curative intent (neoadjuvant, surgery, radiation, and adjuvant treatments) for specific tumor-type and stage per investigator's/primary physician's or research team's judgment. Curative treatment regimens including chemotherapy, radiation, treatment sequencing, and surgery should have been followed as per local standards and NCCN guidelines or non-standard curative-intent therapy through a clinical trial at the discretion of the investigator/treating physician.
6. Patients who have undergone definitive, curative-intent treatment of oligometastatic (synchronous or metachronous) disease with NED per investigator judgement are acceptable for enrollment.
7. Must have disease-free status documented by complete physical examination and imaging studies with no evidence of recurrent, residual, or metastatic disease on standard imaging (chest, abdomen, and pelvis captured by CT chest and CT or MRI of abdomen and pelvis) per investigator assessment within 28 days prior to enrollment
8. Must have a tumor-specific ctDNA SignateraTM test with a positive result (any mean tumor molecule/mL) drawn within 1 year of completing all curative-intent treatment and within 28 days prior to enrollment. In the setting of a negative scan for recurrence, this will be defined as subclinical molecular disease.
9. ECOG Performance Status of 0-2
10. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 28 days prior to initiation of study treatment:

    * ANC ≥1.5 x 109/L (1500/uL) without granulocyte colony-stimulating factor support
    * Lymphocyte count ≥ 0.5 x 10^9/L (500/uL)
    * Platelet count ≥ 75 x 10^9/L (75,000/uL) without transfusion
    * Hemoglobin ≥ 90 g/L (9 g/dL) Patients may be transfused to meet this criterion.
    * AST, ALT, and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN)
    * Note: for HCC, AST, ALT, and alkaline phosphatase (ALP) ≤ 5 x upper limit of normal (ULN)
    * Serum bilirubin ≤ 1.5 x ULN with the following exception: Patients with known Gilbert disease or HCC: serum bilirubin ≤3 x ULN
    * Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
    * Urine dipstick for proteinuria < 2 + (if ≥ 2+ proteinuria on dipstick urinalysis, patient should undergo 24-hour urine collection and must demonstrate < 1 g protein in 24 hours).
    * Serum albumin ≥ 25 g/L (2.5 g/dL). Cut-off of ≥ 28 g/L (2.8 g/dL) will be used for HCC patients.
    * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN. Note: for HCC patients INR or aPTT should be ≤ 2 x ULN.
11. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
12. Negative HIV test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200µL, and have an undetectable viral load.
13. Select patients with well compensated, treated HBV infection and chronic HCV infection may be considered
14. Women of childbearing potential must have a negative serum test result within 28 days prior to initiation of study treatment. If a urine pregnancy test is positive, it must be confirmed by a serum pregnancy test.
15. Women must not be breastfeeding.
16. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs as defined below: o Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 5 months after the final dose of atezolizumab and for 6 months after the last dose of bevacizumab. o Women must refrain from donating eggs during this same period. o A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
17. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: o With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of bevacizumab. Men must refrain from donating sperm during this same period. o With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of bevacizumab to avoid exposing the embryo. o The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.

Exclusion Criteria:

1. There is suspicion or evidence of gross residual, recurrent, or metastatic disease present on physical exam, imaging, or by biopsy within 28 days of starting study treatment.
2. Patients who were/are eligible for but have not received all guideline-recommended standard of care therapy within the recommended time-frame for definitive treatment. The exception (permitting inclusion) would be if any standard of care treatment was deferred due to valid medical reasoning based on the investigator's discretion or patient's preference.
3. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix 6 for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions: o Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. o Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. o Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: - Rash must cover < 10% of body surface area; - Disease is well controlled at baseline and requires only low-potency topical corticosteroids; - No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
4. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan; History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
5. Active tuberculosis
6. Clinically significant cardiovascular disease, such as cerebrovascular accidents within 12 months prior to randomization, myocardial infarction within 12 months prior to study treatment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with study treatment.
7. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization.
8. Inadequately controlled hypertension (defined as systolic blood pressure >150mmHg and/or diastolic blood pressure >100 mmHg), based on an average of ≥ 3 BP blood pressure readings on ≥ 2 sessions. Anti-hypertensive therapy to achieve these parameters is allowable.
9. History of hypertensive crisis or hypertensive encephalopathy
10. History of Grade ≥ 4 venous thromboembolism
11. History or evidence upon physical or neurological examination of central nervous system bleed
12. History of Grade ≥ 2 hemoptysis (defined as ≥ 2.5 mL of bright red blood per episode) within 1 month prior to screening.
13. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation).
14. Current or recent (<10 days prior to initiation of study treatment) use of aspirin (>325 mg/day), or clopidogrel (>75 mg/day) Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or aPTT is within therapeutic limits (according to institution standards) within 7 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥ 2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. For prophylactic use of anticoagulants or thrombolytic therapies, local label approved dose levels may be used. The use of direct oral anticoagulant therapies such as dabigatran (Pradaxa) and rivaroxaban (Xarelto) is not recommended due to bleeding risk.
15. Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID); o Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or joint pain is allowed.
16. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to initiation of study treatment, or anticipation of need for major surgical procedure during the course of the study.
17. Local therapy to liver or other organ (e.g. radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, transarterial chemoembolization, transarterial embolization, etc.) within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure.
18. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding in high-risk patients (patients with HCC, cirrhosis, or other conditions predisposing patients to high-risks of portal hypertension).
19. High risk patients must undergo an esophagogastroduodenoscopy (EGD) and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months prior to initiation of study treatment do not need to repeat the procedure.
20. A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
21. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of study treatment.
22. Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
23. Active infection requiring IV antibiotics at the time of initiation of study treatment.
24. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
25. History of abdominal fistula, GI perforation, intra-abdominal abscess, or active GI bleeding within 6 months prior to study treatment. o If GI bleeding was from a lesion or a condition that was appropriately treated and patient is deemed to be low risk for recurrent GI bleed per investigator judgement, enrollment will be allowed.
26. Serious, non-healing wound, active ulcer, or untreated bone fracture
27. Subjects with previous malignancies (separate from the malignancy for which patient is being enrolled) are excluded. Exceptions include another malignancy for which a complete remission was achieved at least 5 years prior to study entry and no additional therapy is required or anticipated to be required during the study period. Other exceptions include malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, Stage I uterine cancer or others based on the physician/investigator's discretion.
28. Prior allogeneic stem cell or solid organ transplantation
29. Any other disease, active infection, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
30. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
31. Treatment with investigational therapy within 28 days prior to initiation of study treatment
32. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
33. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
34. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: o Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained. o Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
35. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
36. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulation
37. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab or 6 months after the final dose of bevacizumab.

    Women of childbearing potential must have a negative serum or urine pregnancy test result within 28 days prior to initiation of study treatment.
38. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
39. History of leptomeningeal disease
40. Uncontrolled tumor-related pain
41. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently); Patients with indwelling catheters (e.g., PleurX) are allowed.
42. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. Brain scans are not required to be performed at screening but can be done at the clinician's or investigator's discretion depending on clinical history. Asymptomatic patients with previous definitively (with curative-intent) treated CNS lesions that are believed to have no evidence of residual disease per investigator judgement are eligible, provided that all of the following criteria are met: - The patient has no history of intracranial hemorrhage or spinal cord hemorrhage; - The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.; - The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. - If the patient is receiving anti-convulsant therapy, the dose is considered stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rates of SignateraTM ctDNA positive Patient identification | 12 months
  The number of local and regional SignateraTM ctDNA positive patients identified over 12 months in the setting of NED after all SOC definitive therapies (identified patients). This data will be obtained on a local and regional level through the SignateraTM company, Natera.
Rate of Enrollment | 12 months
  Percentage and absolute number of contacted patients who ultimately enrolled on trial (enrolled patients)
Rate of ctDNA Complete Response (CR) | 12 weeks from start of treatment
  Percentage of patients in each cohort (and collectively) who achieve ctDNA CR (defined as ctDNA clearance on two sequential tests compared to baseline ctDNA and ongoing NED clinically/radiographically) within 12 weeks ± 14 days of study therapy.
Rate of ctDNA Partial Response (PR) | 12 weeks from start of treatment
  Percentage of patients in each cohort (and collectively) who achieve ctDNA PR (ctDNA does not clear on two sequential tests, ctDNA does not double on each of two consecutive tests, does not increase on each of three consecutive tests, and ongoing NED clinically/radiographically) within 12 weeks ± 14 days of study therapy.
Rate of ctDNA Progression of Disease (POD) or Clinical/radiographic Relapse | 12 weeks from start of treatment
  Rate of ctDNA POD or clinical/radiographic relapse is defined as the percentage of patients in each cohort (and collectively) who experience ctDNA doubling (at least) on each of two consecutive, sequential tests using the prior ctDNA value as the reference point for doubling for each test, ctDNA rise on each of three consecutive ctDNA tests using the prior ctDNA value as the reference point for each test (ctDNA POD), or clinical/radiographic relapse within 12 weeks ± 14 days of study therapy.

SECONDARY OUTCOMES:
Toxicity by CTCAE v5.0 criteria | 12 months
  Toxicity and safety analysis will occur in patients who received at least one full or partial dose of study treatment. Adverse events will be graded per NCI CTCAE v.5.0.
Reasons for failure of enrollment | 12 months
  Reasons for failure of enrollment characterized as patient preference, physician preference, or ineligibility, among others of identified and contacted patients will be reported

CONTACTS AND LOCATIONS:
Overall Officials: John L. Marshall, MD, Principal Investigator — Georgetown University
Locations (3):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey